CLINICAL TRIAL: NCT07151547
Title: Determination of Cut-Off Values for Gait Variability and Balance Scores in Patients With Multiple Sclerosis
Brief Title: Cut-Off Values for Gait and Balance in MS
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Other Study IDs: Gait Variability
Record Dates: First submitted 2025-08-06; First posted 2025-09-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: cut-off; falls; gait variability; limits of stability; postural sways; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: • Patients diagnosed with MS by a neurologist according to the McDonald criteria, aged 18 years or older, having an EDSS score of ≤ 5 (able to walk independently), and having a Mini-Mental State Examination score of 24 or higher will be included in the study.

SUMMARY:
Purpose of the Study:

The aim of this study is to determine the cut-off values of gait variability and limits of stability-postural sways scores in patients with MS in order to identify fall risk at an early stage and take necessary precautions. Additionally, the study aims to compare the effectiveness of these parameters in distinguishing between fallers and non-fallers.

The study includes four hypotheses:

H₁: Gait variability scores can differentiate between fallers and non-fallers in patients with MS.

H₂: Limits of stability and postural sways scores can differentiate between fallers and non-fallers in patients with MS.

H₃: Gait variability scores provide higher sensitivity and specificity than stability limits and postural sway scores in distinguishing between fallers and non-fallers in patients with MS.

H₄: Limits of stability and postural sways scores provide higher sensitivity and specificity than gait variability scores in distinguishing between fallers and non-fallers in patients with MS.

DETAILED DESCRIPTION:
Gait variability will be assessed using the GaitRite gait analysis system. Limits of stability and postural sways will be evaluated using the Bertec Balance Check Screener™ force platform system. Patients' fall history (number of falls, fear of falling, location of falls, presence of injury, etc.) will also be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS by a neurologist according to the McDonald criteria
* Aged 18 years or older
* EDSS ≤ 5 (able to walk independently)
* Mini-Mental State Examination score of 24 or higher

Exclusion Criteria:

* Patients with neurological conditions other than MS that may affect independent walking or standing, those with lower extremity pain, or a history of lower extremity fractures within the past 6 months
* Patients who do not agree to participate or do not provide written informed consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients with the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Limits of Stability | up to 5 months
  Limits of stability assessment will be conducted using the Bertec Balance Check Screener™ force platform system (45×45 cm, 13 cm thick), which detects body movements via foot pressure.Limits of stability will be measured by asking participants to lean maximally in four directions (forward, backward, right, left) without losing balance. Stability scores (in cm and %) will be calculated using Balance Check Software.
Postural sways | up to 5 months
  Postural sways assessment will be conducted using the Bertec Balance Check Screener™ force platform system (45×45 cm, 13 cm thick), which detects body movements via foot pressure. A foam pad of the same size is used to assess postural sway.
  Postural sways will be evaluated under four conditions (eyes open/closed on firm/foam surfaces). Participants will stand still for 10 seconds per condition, repeated three times. The average stability score (%) will be recorded for each condition.
Gait variability | up to 5 months
  Gait variability will be performed using the GAITRite® system, a 4.6-meter portable walkway mat embedded with pressure sensors that record step data without interfering with the natural gait. Participants will walk naturally across the mat three times; the average of the trials will be analyzed. Gait variability will be expressed as the coefficient of variation (CV) (%).
  Using this formula:
  CV (%) = (standard deviation/mean) × 100.
Fall Histories | up to 5 months
  The following fall-related information will be recorded:
  Number of Falls
  Cause of Fall
  Time of Fall
  Activity During Which the Fall Occurred
  Type of Fall
  Fall-Related Injury / If Present, Type of Injury

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Kılınç, Principal Investigator — Hacettepe University; Ender Ayvat, Principal Investigator — Hacettepe University; Fatma Ayvat, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)